CLINICAL TRIAL: NCT00365248
Title: A Prospective, Multi-centre Phase III-b Study of TachoSil in Paediatric Patients Scheduled for Resection of the Liver With or Without Segmental Liver Transplantation.
Brief Title: TachoSil Paediatric Liver Trial (TC-019-IN)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Nycomed (Industry)
Responsible Party: Nycomed, Nycomed
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TC-019-IN; 2004-005028-42
Record Dates: First submitted 2006-08-16; First posted 2006-08-17 (Estimated); Last update posted 2012-05-07 (Estimated); Status verified 2008-07

CONDITIONS: Liver Diseases
Keywords: Surgical resection of the liver with or without segmental transplantation
MeSH Terms: conditions — Liver Diseases | interventions — Fibrinogen; TachoSil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Fibrinogen human (TachoSil) — Resection of the liver with or without segmental liver transplantation

SUMMARY:
The overall objective is to assess the haemostatic efficacy and safety of TachoSil for control of local bleeding in paediatric patients undergoing surgical resection of the liver with our without segmental liver transplantation.

ELIGIBILITY:
Inclusion criteria:

1. Has the parent(s)/legal guardian given informed consent according to local requirements before any trial related activities?
2. Is the child above 4 weeks and below 6 years of age?
3. Has at least segmental resection (anatomical/non-anatomical) of the liver and primary haemostatic treatment been performed? or Has resection of the liver and placement of a segmental liver graft and primary haemostatic treatment been performed?
4. Is only minor, i.e. oozing, or moderate haemorrhage persisting after primary surgical haemostatic procedures of the major vessels (no pulsating arterial haemorrhage and/or major venous bleeding)?

All inclusion criteria must be answered "yes" for a child to participate in the study.

Exclusion criteria:

1. Was the child retransplanted or had liver transplantation in combination with other organs?
2. Was there anamnestic or laboratory evidence of congenital coagulation disorders including Haemophilia A or B and von Willebrand disease?
3. Has the child a history of allergic reactions after application of human fibrinogen, human thrombin and/or collagen of any origin?
4. Has the child fulminant hepatic failure, portal vein thrombosis or anamnestic or clinical evidence of cirrhotic condition of the liver, including cirrhosis due to genetic deficiency of a1 - Antitrypsin?
5. Did the child undergo an emergency operation?
6. Does the child participate in another clinical trial during the intra-operative phase?
7. Has any serious surgical complication occurred?
8. Has any fibrin glue haemostatic (including TachoSil ® ) been used on the target wound before the planned application of TachoSil ® ? To participate in the study all exclusion criteria must be answered "No" for a child having segmental resection. For a child having total hepatectomy and placement of a segmental liver transplant criteria 4 and 5 can be answered "Yes".

Ages: 4 Weeks to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 16 (Actual)
Dates: Start 2005-10; Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
The primary objective is to collect data on efficacy, i.e. intra-operative haemostasis, and safety of TachoSil ® as treatment to control local bleeding in children undergoing surgical resection of the liver with or without segmental transplantation. | 7½ months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Operations, Study Chair — Headquaters
Locations (1):
- Nycomed, Roskilde, Denmark